CLINICAL TRIAL: NCT05192031
Title: Implementation of Smoking Cessation Support During Lung Cancer Workup: a Pragmatic, Cluster-randomised Controlled Trial and an Interview-based Study of Patients' and Healthcare Professionals' Experiences
Brief Title: Implementation of Smoking Cessation Support During Lung Cancer Workup
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Naestved Hospital (Other); Odense University Hospital (Other); Zealand University Hospital (Other); Bispebjerg Hospital (Other); Hospital of Southern Jutland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: START
Record Dates: First submitted 2021-12-17; First posted 2022-01-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Suspected Lung Cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking cessation support (Experimental)
  Interventions: Behavioral: Smoking cessation support
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Smoking cessation support — Training healthcare professionals to deliver smoking cessation support as part of hospital-based lung cancer workup.
  Arms: Smoking cessation support

SUMMARY:
The aim of the present project is to implement smoking cessation support in hospital-based lung cancer workup. The effect on 1) patients' smoking cessation attempts, motivation, quality of life and psychosocial consequences of lung cancer workup as well as 2) hospitals' number of referrals to municipality-based smoking cessation programmes will be evaluated in a pragmatic, cluster-randomised controlled setup, where participating hospitals will be assigned to the intervention arm (implementation of smoking cessation support) or the control arm (usual practice). Patients' and healthcare professionals' experiences with and barriers towards smoking cessation support will be explored in an interview-based, qualitative study.

ELIGIBILITY:
Inclusion Criteria:

* Referred to lung cancer workup at participating hospital
* Able to speak and understand Danish

Exclusion Criteria:

* Unable to complete electronic questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients making an attempt at smoking cessation during lung cancer workup | 6 weeks after baseline
  Binary outcome (Attempt: yes, no)

SECONDARY OUTCOMES:
Motivation to quit smoking | 6 weeks, 3, 6, and 12 months after baseline
  Numeric rating scale (0-10) with higher score indicating stronger motivation
Proportion of patients who are not smoking at the time of measurement | 6 weeks, 3, 6, and 12 months after baseline
  Binary outcome (Currently smoking: yes, no)
Quality of life as measured by the 36 item Short Form Survey (SF-36) | 6 weeks, 3, 6, and 12 months after baseline
  SF-36, two components: Mental and Physical. Each components scale has a total score range from 5 (worst health) to 80 (best health)
Psychosocial consequences of lung cancer workup | 6 weeks after baseline
  Consequences of Screening - Lung Cancer Questionnaire (adapted to the lung cancer workup setting). Items in Part 1 of the questionnaire focuses on experiences during the cancer workup with a total score range from 0 (low level of psychosocial consequences) to 72 (high level of psychosocial consequences). Items in Part 2 of the questionnaire focuses on experiences after the cancer workup with a total score range from 0 (low level of psychosocial consequences) to 22 (high level of psychosocial consequences).
Hospitals' number of referrals to municipality-based smoking cessation programmes | Change from one year before to one year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anders Løkke, MD, Study Director — Vejle Hospital, Lillebaelt Hospital; Ole Hilberg, Prof, Study Director — Vejle Hospital, Lillebaelt Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No